CLINICAL TRIAL: NCT06223971
Title: A Phase l Study to Assess the Safety and Tolerability of PET Imaging With [11 C]CPPC [5-cyano-N-( 4-( 4-[l l CJ me1hylpiperazin-l-yl)-2-(Piperidin-l-yl)Phenyl)Furan-2-carboxamide] Radioligand and Magnetic Resonance (MR) Imaging in Patients With Long COVID.
Brief Title: Long COVID-19 [11C]CPPC Study
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00361674
Record Dates: First submitted 2024-01-23; First posted 2024-01-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: COVID Long-Haul
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients with history of COVID-19 infection and still experiencing symptoms (Long-COVID) (Experimental): Participants with a diagnosis of Long- COVID will receive a single dose of [11C]CPPC (370 megabecquerel (MBq) (X±1 mCi)) intravenously and subsequent positron emission tomography (PET) scan.
  Interventions: Drug: [11C]CPPC Injection
- Healthy Participants with history of COVID-19 infection but not experiencing any symptoms. (Experimental): Healthy participants (without any history of post-COVID symptoms) will receive a single dose of [11C]CPPC (370 megabecquerel (MBq) (X±1 mCi)) intravenously and subsequent positron emission tomography (PET) scan.
  Interventions: Drug: [11C]CPPC Injection

INTERVENTIONS:
Drug: [11C]CPPC Injection — A single dose of [11C]CPPC (370 megabecquerel (MBq) (X±1 mCi)) intravenously and subsequent positron emission tomography (PET) scan.
  Other Name: [5-cyano-N-(4-(4-[11C]methylpiperazin-1-yl)-2-(piperidin-1-yl)phenyl)furan-2-carboxamide]
  Arms: Patients with history of COVID-19 infection and still experiencing symptoms (Long-COVID)
Drug: [11C]CPPC Injection — A single dose of [11C]CPPC (370 megabecquerel (MBq) (X±1 mCi)) intravenously and subsequent positron emission tomography (PET) scan.
  Other Name: [5-cyano-N-(4-(4-[11C]methylpiperazin-1-yl)-2-(piperidin-1-yl)phenyl)furan-2-carboxamide]
  Arms: Healthy Participants with history of COVID-19 infection but not experiencing any symptoms.

SUMMARY:
The goal of this study is to evaluate the safety of using the [5-cyano-N-(4-(4-[11C]Methylpiperazin-1-yl)-2-(Piperidin-1-yl)Phenyl)Furan-2-carboxamide] ([11C]CPPC) radiotracer in positron emission tomography (PET) imaging of people with history of COVID-19 infection, with and without symptoms. The investigators are also interested to see whether use of this radiotracer reveals imaging differences between patients with history of COVID-19 infection and still exhibiting symptoms or healthy patients with history of COVID-19 infection but exhibiting no current symptoms.

DETAILED DESCRIPTION:
This is a Phase 1 study of safety and tolerability of an investigational radiotracer drug called [5-cyano-N-(4-(4-[11C]Methylpiperazin-1-yl)-2-(Piperidin-1-yl)Phenyl)Furan-2-carboxamide] ([11C]CPPC). A radiotracer is a substance that chemically marks certain structures in the body. In this case, [11C]CPPC highlights structures expressing colony stimulating factor receptor (CSF1R), a receptor that is expressed on microglial cells. A safety and tolerability study is looking to see if there are any unanticipated, possibly harmful, effects of the use of the radiotracer in humans. However, ultimately, the investigators would like to know if this drug can be used to make better images of the brain for patients with history of COVID-19 infection, which could help doctors better understand the disease and help take care of patients suffering from Long COVID symptoms. This study will use a radiotracer to look for a chemical receptor which may be affected in patients who report of Long COVID. After receiving the radiotracer, participants' brains will be scanned with a positron emission tomography (PET) imaging machine. Each participant will also undergo magnetic resonance imaging (MRI) without contrast, detailed cognitive testing and a neurological exam. This study will assess possible associations between COVID-19 infection, cognitive function, other neurological symptoms, and 11C-CPPC PET neuroimaging in subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand the requirements of the study, provide written informed consent, understand and provide written authorization for the use and disclosure of Protected Health Information (PHI) [per Health Insurance Portability and Accountability Act (HIPAA) Privacy Ruling] and comply with the study procedures.
2. Documented history of COVID infection at least 6 - 12 months before enrollment.
3. Men and women at least 18 years old.
4. Women must have a negative serum pregnancy test and practice an acceptable method of contraception or be of non-childbearing potential (post-menopausal for at least 2 years or who have undergone hysterectomy, oophorectomy or surgical sterilization).
5. Geographic accessibility to the study center and the ability to travel to the clinic for study visits.
6. Agrees to the visit schedule as outlined in the informed consent.
7. Pre-study labs within normal range, or if abnormal, deemed not clinically significant by the site investigator.

Exclusion Criteria:

1. History of recent nosocomial infection.
2. History of chronic neurological disorder, such as epilepsy, or structural Central Nervous System (CNS) abnormality such as stroke or arteriovenous malformation.
3. History of head trauma with prolonged loss of consciousness (>10 minutes) or any neurological condition including stroke, seizure (excluding childhood febrile seizure), or visible structural abnormality on prior MRI.
4. Active or recent (in the past year) substance dependence (drugs-including nicotine, marijuana or alcohol).
5. Receipt of any investigational drug, device or biologic within 30 days of administration of study compound.
6. Use of anti-inflammatory medications, immunosuppressants, or benzodiazepines within 7 days of administration of study compound.
7. Any concomitant medical disease or condition limiting the safety to participate including, but not limited to:

   * Coagulopathy
   * Active infection
8. Contraindications to MRI scanning to include pacemakers, metallic implants/prosthesis or prohibitive claustrophobia, etc.
9. Contraindications to PET scanning to include pregnancy, etc.
10. Any medical condition that in the opinion of the study investigators would constitute a safety risk to the subject.
11. Any radiation exposure in the past calendar year that in combination with the radiation exposure from this study would exceed 5 rem.
12. Any history of learning disability or special education (due to the potential to affect performance on neuropsychological testing).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of one dose level of [11C]CPPC when administered intravenously. | Baseline and up to 2 days follow-up after scan
  Safety and tolerability will be determined by evaluation of spontaneously reported adverse events, clinical laboratory test results, physical, cognitive and neurologic exams and imaging (PET).
Safety of use of [11C]CPPC in patients with Long-COVID and healthy participants with history of COVID-19 infection as assessed by a change in complete blood count (CBC) test. | Baseline and up to 2 days follow-up after scan
  Safety of use of [11C]CPPC in positron emission tomography (PET) neuroimaging of patients with Long-Covid and healthy participants with history of COVID-19 infection. Safety will be assessed by monitoring of the complete blood count (CBC) for a change from baseline that is outside of the normal range.
Safety of use of [11C]CPPC in patients with Long-COVID and healthy participants with history of COVID-19 infection as assessed by a change in complete metabolic panel (CMP) test. | Baseline and up to 2 days follow-up after scan
  Safety of use of [11C]CPPC in positron emission tomography (PET) neuroimaging of patients with Long-COVID and healthy participants with history of COVID-19 infection. Safety will be assessed by a change in the CMP from baseline that is outside of the normal range

SECONDARY OUTCOMES:
Biodistribution of [11C]CPPC by PET imaging | 1 day
  Image analysis of PET imaging obtained of patients and healthy participants. The PET compartmental model fits will be applied to the regional time activity curves (TACs) will be first assessed visually before the relative goodness of fit will be assessed using the statistical F test.
Cognitive function as assessed by the NIH Toolbox Cognition Battery (NIHTB-CB) | 1 day
  NIH Toolbox Cognition Battery (NIHTB-CB), which is an iPad-based instrument assessing five cognitive sub-domains: Language, Executive Function, Episodic Memory, Processing Speed, and Working Memory. Score range 59 - 140, higher score means better cognition.
Neuro-psychological assessment as assessed by the The Rey-Osterrieth complex figure test (ROCF) | 1 day
  The Rey-Osterrieth complex figure test (ROCF) is a neuro-psychological assessment in which participants are asked to reproduce a complicated line drawing, first by copying it freehand (recognition), and then drawing from memory (recall). Scoring of drawings is based on the 36-point scoring system (0 being the worst score and 36 the best).
Global cognitive function as assessed by the Mini-Mental State Exam (MMSE) | 1 day
  The MMSE is a measure of global cognitive function, scores range from 0-30, a lower score indicates greater cognitive impairment.
Dementia as assessed by the Clinical Dementia Rating (CDR) scale | 1 day
  The Clinical Dementia Rating Dementia Staging Instrument minimum score = 0, maximum score = 18. Low scores indicate less problems.
Hospital Anxiety and Depression Scale (HADS) score | 1 day
  Scoring for the Hospital Anxiety and Depression scale is 0-21; Normal (0-7); Borderline Abnormal Case (8-10); and Abnormal Case (11-21) higher score indicates worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Licia Luna, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No